CLINICAL TRIAL: NCT04589481
Title: Effectiveness of Different Candies Against Bad Breath
Acronym: HALIDROP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Ricola Group AG Schweiz (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2020-01943; ex20Filippi
Record Dates: First submitted 2020-10-14; First posted 2020-10-19 (Actual); Last update posted 2021-06-02 (Actual); Status verified 2021-06

CONDITIONS: Bad Breath
Keywords: halitosis; volatile sulphur compounds
MeSH Terms: conditions — Halitosis

STUDY DESIGN:
Intervention Model Description: Three different variants of a candy are being tested by each participant. The candies are randomly assigned to the subjects, so that each subject has tested each of the three candies once. Randomization creates a different order for each participant. The study will be carried out on three different days.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- candy intake (Experimental)
  Interventions: Other: Intake of 3 different candies against bad breath

INTERVENTIONS:
Other: Intake of 3 different candies against bad breath — Intake of 3 different candies against bad breath on three different days (2-days interval each) after artificially creating a temporary bad breath (by eating of chips and cheese); analysis of breathing during intake of candy both subjectively and objectively

SUMMARY:
This study is to analyze whether the candies can relieve or eliminate bad breath, both subjectively and objectively.

DETAILED DESCRIPTION:
This study is to systematically examine an existing candy, which is easily available and is intended to relieve or eliminate bad breath. The main aim of the study is to determine the effectiveness of the candies on the subjective perception of bad breath. The secondary outcome of the study is to investigate whether there is actually a decrease in volatile sulphur compounds (VSC) in the exhaled air and also a decrease in bad breath during organoleptic measurement.

The purpose of the study is to investigate whether the different candies can relieve or eliminate bad breath, both subjectively and objectively.

ELIGIBILITY:
Inclusion Criteria:

* Non- smoker
* No general medical illness or medication

Exclusion Criteria:

* Allergies/intolerances to ingredients of the products used
* Chronic diseases
* Smoker
* Pregnancy

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2021-02-23 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
Organoleptic analysis of breathing air sample | max 60 minutes at 3 different days
  Assessment of the patient's bad breath on the basis of the subjective assessment of an investigator (scale of 0 to 5 (0, no odor; 1, questionable odor; 2, slight malodor; 3, moderate malodor; 4, strong malodor; 5, severe malodor))
Measurement of volatile sulphur compounds (VSC) in ppb (parts per billion). | max 60 minutes at 3 different days
  Assessment of the patient's bad breath on the basis of the objective assessment by a sulfide monitor (HaliSens® AI Analytical Innovations GmbH, Moosbach, Germany)

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Filippi, Prof. Dr. med. dent., Principal Investigator — Universitäres Zentrum für Zahnmedizin Basel (UZB)
Locations (1):
- Universitäres Zentrum für Zahnmedizin UZB, Basel, Switzerland